CLINICAL TRIAL: NCT01613950
Title: A Phase IB, Multicenter, Open-label Dose Escalation Study of the PI3K Inhibitor BYL719 in Combination With the HSP90 Inhibitor AUY922 in Patients With Advanced or Metastatic Gastric Cancer Carrying a Molecular Alteration of PIK3CA or an Amplification of HER2
Brief Title: PI3K Inhibitor BYL719 in Combination With the HSP90 Inhibitor AUY922 in Patients With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X2103; 2011-005978-40 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-07 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2017-02

CONDITIONS: Stomach Neoplasms Esophageal Neoplasms Metastatic Gastric Cancer Mutated PI3KCA Protein Overexpressed HER2 Protein
Keywords: gastric cancer advanced gastric or metastatic gastric cancer PI3K PIK3CA mutation Her2 amplification HSP90 inhibitor PI3K inhibitor PIK3CA amplification
MeSH Terms: interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Alpelisib

ARMS (1):
- BYL719 + AUY922 (Experimental): Dose finding study to estimate the maximum tolerated dose(s) (MTD) and/or recommended dose(s) for safety expansion (RDE) followed by an expansion phase to further assess the safety and preliminary activity of the combination. BYL719 tablets will be administered orally on a daily schedule (q.d.). a b.i.d. regimen may be explored. AUY922 will be administered by IV infusion once per week.
  Interventions: Drug: AUY922; Drug: BYL719

INTERVENTIONS:
Drug: AUY922 — AUY922 is a non-geldanamycin inhibitor of the heat shock protein 90 (HSP90).
Drug: BYL719 — BYL719 is an oral α-specific phosphatidylinositol-3-kinase (PI3K) inhibitor.

SUMMARY:
The study is intended to investigate the safety of BYL719 and AUY922 in patients with advanced gastric cancer, and to determine the MTD and/or RDE of both drugs in combination. In addition, the preliminary efficacy of BYL719 in combination with AUY922, and the pharmacokinetics of both drugs will be assessed. Patients will be eligible for this study, if their tumors carry either a molecular alteration of PIK3CA, or an amplification of HER2.

The study includes a dose escalation part followed by a safety expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction;
* Patients must not have a complete gastrectomy;
* gastric tumors carrying PIK3CA mutation or amplification, or HER2-overexpression, or both;
* at least one but no more than three previous lines of treatment for advanced or metastatic disease;
* Patients with PIK3CA mutated or amplified tumors must have failed at least one line but no more than three lines of standard chemotherapy and/or targeted agents;Patients with HER2 amplified tumor must have failed at least one line, but no more than three lines, with or without anti-HER2 therapy. All HER2 positive patients are expected to have received trastuzumab unless contraindications were present or trastuzumab was unavailable;
* Performance Status (PS) ≤ 1 ;
* Adequate bone marrow, liver and other organ functions and laboratory parameters;
* Recovery from all AEs of previous anti-cancer therapies, including surgery and radiotherapy, to baseline or to CTCAE Grade ≤ 1, except for alopecia;Negative serum pregnancy (β hCG) test within 72 hrs before starting study treatment in all pre-menopausal women and women < 12 months after the onset of menopause.

  * Exclusion Criteria:
* Progressive disease during or after prior combination treatment with PI3K-inhibitors and HSP90- inhibitors;
* history of prior significant toxicity from another PI3K- or HSP90- inhibitor requiring discontinuation of treatment;
* primary CNS tumor or uncontrolled CNS metastasest;
* Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment;
* Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with fasting glucose ≥ 140 mg/dL / 7.8 mmol/L, history of clinically significant gestational diabetes mellitus or documented steroid-induced diabetes mellitus;Patients with diarrhea CTCAE Grade ≥ 2 ;
* Patients with acute or chronic pancreatitis; History or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or ophthalmopathy as assessed by ophthalmologic examination at baseline that would be considered a risk factor for CSR/RVO;
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719;
* Patients receiving chronic slow-release formulation of Proton Pump Inhibitors (PPI), H2-antagonists or other gastric pH elevating agents;
* Treatment with therapeutic doses of coumarin-based anticoagulants (e.g., warfarin sodium, Coumadin®). Low doses of courmarin-based anticoagulants;
* Patients receiving chronic or high dose corticosteroids therapy; other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicities. | cycle 1
  To determine the maximum tolerated dose (MTD) and/or Recommended dose for expansion (RDE) and schedule of BYL719 and AUY922 when used as a combination in patients with advanced or metastatic gastric cancer carrying a molecular alteration of PIK3CA and/or an amplification of HER2. 1 cycle = 28days

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | duration of the study, an expected average of 24 months
  To characterize the safety and tolerability of BYL719 and AUY922 in combination.
Best Overall Response (BOR) as per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 | every 6 weeks
  To assess the preliminary anti-tumor activity of BYL719/AUY922 combination from Treatment start to disease progression
Plasma concentration versus time profiles of BYL719 as single agent an in combination with AUY922. | 2 months
  To determine the single dose PK of BYL719 single dose, and multiple doses PK of BYL719.
Overall response rate (ORR) as per RECIST version 1.1 | an expected average of 12 months
  To assess the preliminary anti-tumor activity of BYL719/AUY922 combination.
Progression free survival (PFS) as per RECIST version 1.1 | every 6 weeks
  To assess the preliminary anti-tumor activity of BYL719/AUY922 combination.
Overall survival (OS) | approximately 1 year
  To assess the preliminary anti-tumor activity of BYL719/AUY922 combination.
Overall survival rate at 6 months (OS6) | 6 months
  To assess the preliminary anti-tumor activity of BYL719/AUY922 combination.
Frequency and severity of serious adverse events (SAEs) | duration of the study, an expected average of 24 months
  To characterize the safety and tolerability of BYL719 and AUY922 in combination.
Plasma concentration versus time profile of AUY922 as single agent and in combination with BYL719 | 2 months
  To determine the single dose and multiple dose pharmacokinetics of AUY922
Plasma concentration versus time profile of the AUY922 metabolite BJP762 | 2 months
  To determine pharmacokinetics of BJP762 after single dose and multiple dose of AUY922
Severity of adverse events (AEs) | duration of the study, an expected average of 24 months
  To characterize the safety and tolerability of BYL719 and AUY922 in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - Massachusetts General Hospital Mass General 2, Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center Gastrointestinal Med. Oncology, Houston, Texas
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Chuo-ku, Tokyo, Japan
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Bellinzona, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

REFERENCES:
- See also: Results for CBYL719X2103 can be found on the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13567